CLINICAL TRIAL: NCT06079658
Title: The Effects of Continuous vs. Intermittent Caloric Restriction on Fat Loss: A Randomized Controlled Trial
Brief Title: The Effects of Continuous vs. Intermittent Caloric Restriction on Fat Los
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coastal Carolina University (Other)
Responsible Party: Principal Investigator, Kelly Johnson, Assistant Professor Exercise Science, Coastal Carolina University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.06
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Weight Loss, Telehealth, health Coaching, Diet Breaks
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: All participants were randomized in a balanced fashion and stratified by body fat percentage into either one of the two intervention groups.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Caloric Restriction (CCR) group: (Experimental): Participants in this group will be placed on a diet that is prescribed a 25% reduction from maintenance calories (calories to maintain current body weight) with a dietary protein intake of 1.2 g of protein/kg body mass and remaining calories split evenly between fat and carbohydrate. In this group they will adhere to a 25% caloric reduction daily for 12 weeks.
  Interventions: Behavioral: Continuous Caloric Restriction versus Intermittent Caloric Restriction on Fat Loss
- Intermittent Caloric Restriction (ICR) group: (Experimental): Participants in this group will be placed on a diet that is prescribed a 25% reduction from maintenance calories (calories to maintain current body weight) with a dietary protein intake of 1.2 g of protein/kg body mass and remaining calories split evenly between fat and carbohydrate. Participants will adhere to a 25% caloric deficit daily and on every 7th day they will eat their maintenance calories known as a "diet refeed" and then on the 3rd week they will take a "diet break" of eating their Maintenance calories for 7 days.
  Interventions: Behavioral: Continuous Caloric Restriction versus Intermittent Caloric Restriction on Fat Loss

INTERVENTIONS:
Behavioral: Continuous Caloric Restriction versus Intermittent Caloric Restriction on Fat Loss — This intervention seeks to investigate two different caloric restriction protocol on fat mass.

SUMMARY:
The purpose of this research study examines fat mass loss using a continuous calorie reduction protocol versus continuous caloric restriction interspersed with "diet refeeds" and "diet breaks" over 12 weeks.

DETAILED DESCRIPTION:
In order to lose weight, an individual must sustain an energy deficit (whereby caloric intake is significantly lower than expenditure) over time. However, a rich base of evidence suggests that weight loss often results in a decreased metabolic rate. This decrease, likely the result of a number of physiological and behavioral mechanisms, makes the continuation of weight loss more difficult as well as increases the likelihood of weight regain, or the "rebound" effect (1, 2). One proposed method of promoting the retention of a higher metabolic rate through a period of caloric restriction, and therefore preventing the regain of excess weight after energy restriction is discontinued, is the use of intermittent rather than continuous caloric restriction. Intermittent energy restriction (IER) involves undulating one's energy intake throughout a dieting period as opposed to sustaining a continuous energy deficit.

Research in overweight and obese individuals has shown that periods of moderate caloric restriction interspersed with periods of consuming a diet in balance with one's daily energy needs (caloric maintenance) is at least comparable to continuous energy restriction in terms of weight and fat loss outcomes (3) and may even bestow unique benefits by promoting greater retention of fat-free mass and a higher metabolic rate (4). However, to date, no published research has examined continuous caloric restriction compared to Intermittent energy restriction (diet breaks and diet refeeds) in females only with Obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years of age, 2) Females only, 3) All ethnicities 4). Must reside in Horry County, South Carolina, 5) have a BMI of > 30-45 kg/m2 6) weight stable for the last 3 months 7). Exercise less than 150 minutes of physical activity per week) 8. Have access to an Apple® iPhone or Android® smart phone.

Exclusion Criteria:

* Adults who are physically active greater than 150 minutes per week, participants who were unwilling or unable to attend testing sessions between 6 am and 12 pm, participants planning to take holidays and/or work-related travel during the study period (challenges adherence to the diet, and interferes with testing session scheduling, participants who have lost greater than 10 pounds in the last 3 months, participants has stated an immunodeficiency disorder, kidney disease, heart attack within the last 3 months, has known dementia, brain cancer, current eating disorders, history of significant neurological or psychiatric disorder or any other psychological condition impacting their decision making, currently taking dietary supplements that could profoundly modify metabolism or body weight, has undergone major surgery, less than 4 weeks prior to enrollment in the study, undergone bariatric surgery <12 months prior to starting the study, or diagnosis of type 1 diabetes. Although not anticipated for this study population, women cannot be or suspect they may be pregnant.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Fat Loss | Change in fat mass between baseline (week 0) and post intervention (week 12)
  Investigators examined body composition fat loss between groups baseline (week 0) and post intervention (week 12).

SECONDARY OUTCOMES:
% Weight Loss | Change in % weightloss between baseline (week 0) and post intervention (week 12)
  Investigators examined % body weight loss between groups baseline (week 0) and post intervention (week 12).

CONTACTS AND LOCATIONS:
Locations (1):
- Williams Brice Building, Conway, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trexler ET, Smith-Ryan AE, Norton LE. Metabolic adaptation to weight loss: implications for the athlete. J Int Soc Sports Nutr. 2014 Feb 27;11(1):7. doi: 10.1186/1550-2783-11-7. PMID 24571926
- [Result] Fothergill E, Guo J, Howard L, Kerns JC, Knuth ND, Brychta R, Chen KY, Skarulis MC, Walter M, Walter PJ, Hall KD. Persistent metabolic adaptation 6 years after "The Biggest Loser" competition. Obesity (Silver Spring). 2016 Aug;24(8):1612-9. doi: 10.1002/oby.21538. Epub 2016 May 2. PMID 27136388
- [Result] Arguin H, Dionne IJ, Senechal M, Bouchard DR, Carpentier AC, Ardilouze JL, Tremblay A, Leblanc C, Brochu M. Short- and long-term effects of continuous versus intermittent restrictive diet approaches on body composition and the metabolic profile in overweight and obese postmenopausal women: a pilot study. Menopause. 2012 Aug;19(8):870-6. doi: 10.1097/gme.0b013e318250a287. PMID 22735163
- [Result] Byrne NM, Sainsbury A, King NA, Hills AP, Wood RE. Intermittent energy restriction improves weight loss efficiency in obese men: the MATADOR study. Int J Obes (Lond). 2018 Feb;42(2):129-138. doi: 10.1038/ijo.2017.206. Epub 2017 Aug 17. PMID 28925405